CLINICAL TRIAL: NCT00767624
Title: Improving Depression Outcome by Adding Insomnia Therapy to Antidepressants
Brief Title: TRIAD - Treatment of Insomnia and Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Duke University (Other); University of Pittsburgh (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Rachel Manber, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-08132008-1277; MH78924
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Antidepressive Agents; Desensitization, Psychologic; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antidepressant + desensitization (Other): Combined antidepressant medication (determined by an algorithm) plus desensitization therapy
  Interventions: Drug: Antidepressant; Behavioral: Desensitization Therapy for Insomnia
- antidepressant + cognitive behavioral (Other): Combined antidepressant medication (determined by algorithm) plus cognitive behavioral therapy
  Interventions: Drug: Antidepressant; Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Drug: Antidepressant — Possible antidepressants are sertraline, escitalopram, desvenlafaxine, based on past history, response and tolerance
Behavioral: Desensitization Therapy for Insomnia
  Arms: antidepressant + desensitization
Behavioral: Cognitive Behavioral Therapy for Insomnia
  Arms: antidepressant + cognitive behavioral

SUMMARY:
The aim of the proposed three-site study is to increase the rate of full remission from major depressive disorder (MDD) at the end of 16 weeks of treatment for people who experience both major depressive disorder and insomnia.

DETAILED DESCRIPTION:
Participants with major depressive disorder and insomnia who meet all study criteria will receive state-of-the-art antidepressant medications and one of two insomnia therapies. The specific therapy for insomnia will be determined by chance (like a flip of a coin), with an equal chance to receive either cognitive-behavioral therapy for insomnia or desensitization psychotherapy for insomnia. The study physician will select an initial antidepressant medication from a list of three possible medications . If that medication is not helpful, another medication may be tried after 8 weeks or in the event of severe side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for Major Depressive Disorder
2. Between 18 and 75 years of age and adequately fluent in English
3. Meets criteria for an insomnia disorder

Exclusion Criteria:

1. Women who are currently pregnant, breast-feeding, or not using a reliable birth control method.
2. People for whom the antidepressant medication(s) provided in the study is not indicated
3. People who have had minimum adequate trials of (or have not been able to tolerate) all three study medications.
4. People with uncontrolled medical conditions.
5. People with moderate or severe sleep disorders other than insomnia
6. Individuals on a fixed night shift or rotating work schedule that requires a night shift.
7. Patients with a current principal diagnosis of a psychiatric disorder that necessitates treatment that is not offered in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Manber, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spina MA, Bei B, Rajaratnam SW, Krystal A, Edinger JD, Buysse DJ, Thase M, Manber R. Cognitive behavioural therapy for insomnia reduces actigraphy and diary measured sleep discrepancy for individuals with comorbid insomnia and major depressive disorder: A report from the TRIAD study. Sleep Med. 2024 Feb;114:137-144. doi: 10.1016/j.sleep.2023.12.014. Epub 2023 Dec 24. PMID 38183804
- [Derived] Edinger JD, Smith ED, Buysse DJ, Thase M, Krystal AD, Wiskniewski S, Manber R. Objective sleep duration and response to combined pharmacotherapy and cognitive behavioral insomnia therapy among patients with comorbid depression and insomnia: a report from the TRIAD study. J Clin Sleep Med. 2023 Jun 1;19(6):1111-1120. doi: 10.5664/jcsm.10514. PMID 36798983
- [Derived] Asarnow LD, Bei B, Krystal A, Buysse DJ, Thase ME, Edinger JD, Manber R. Circadian Preference as a Moderator of Depression Outcome Following Cognitive Behavioral Therapy for Insomnia Plus Antidepressant Medications: A Report From the TRIAD Study. J Clin Sleep Med. 2019 Apr 15;15(4):573-580. doi: 10.5664/jcsm.7716. PMID 30952216
- [Derived] Bei B, Asarnow LD, Krystal A, Edinger JD, Buysse DJ, Manber R. Treating insomnia in depression: Insomnia related factors predict long-term depression trajectories. J Consult Clin Psychol. 2018 Mar;86(3):282-293. doi: 10.1037/ccp0000282. PMID 29504795
- [Derived] Manber R, Buysse DJ, Edinger J, Krystal A, Luther JF, Wisniewski SR, Trockel M, Kraemer HC, Thase ME. Efficacy of Cognitive-Behavioral Therapy for Insomnia Combined With Antidepressant Pharmacotherapy in Patients With Comorbid Depression and Insomnia: A Randomized Controlled Trial. J Clin Psychiatry. 2016 Oct;77(10):e1316-e1323. doi: 10.4088/JCP.15m10244. PMID 27788313

RESULTS

PARTICIPANT FLOW:
Groups:
- Antidepressant + Desensitization: Combined antidepressant medication (determined by an algorithm) plus desensitization therapy
  Antidepressant: Possible antidepressants are sertraline, escitalopram, desvenlafaxine, based on past history, response and tolerance
  Desensitization Therapy for Insomnia
- Antidepressant + Cognitive Behavioral: Combined antidepressant medication (determined by algorithm) plus cognitive behavioral therapy
  Antidepressant: Possible antidepressants are sertraline, escitalopram, desvenlafaxine, based on past history, response and tolerance
  Cognitive Behavioral Therapy for Insomnia
Period: Overall Study
Arm/Group | Antidepressant + Desensitization | Antidepressant + Cognitive Behavioral
Started | 75 | 75
Completed | 51 | 58
Not Completed | 24 | 17

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant + Desensitization | Antidepressant + Cognitive Behavioral | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.3) | 48.3 (12.7) | 46.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 53 | 110
  Male | 18 | 22 | 40
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28, with larger numbers representing greater severity. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8- 14); moderate insomnia (15-21); and severe insomnia (22-28).
  units on a scale | 18.3 (3.9) | 19.4 (4.3) | 18.9 (4.1)
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — The HRSD is a 17-item semi-structured interview assessing the severity of depression in the past week. Items are rated on a 3 or 5 point scale. The total score is the sum of individual items, yielding a total score ranging from 0 to 52, with larger numbers representing greater severity. The total score is interpreted as follows: absence of depression (0-7); mild depression (8- 16); moderate depression (17-23); and severe depression (24-52).
  units on a scale | 21.5 (3.7) | 21.9 (3.8) | 21.7 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Depression Remission
Description: Depression remission was defined if both a and b below are satisfied
  1. absence of both depressed mood and anhedonia for at least three consecutive weeks
  2. no more than two other diagnostic criterion symptoms of depression met for at least three consecutive weeks
Time Frame: 16 weeks
Measure: Number; unit: percentage of participants in arm
Arm/Group | Antidepressant + Desensitization | Antidepressant + Cognitive Behavioral
Number analyzed (Participants) | 75 | 75
percentage of participants in arm | 36.0 | 43.8

2. Secondary Outcome: Percentage of Participants in Insomnia Remission
Description: Remission was defined as endpoint ISI<8. The ISI scale score ranges from 0 to 28 with lower scores representing less severe insomnia. A score of 0-7 is interpreted as absence of insomnia.
Time Frame: 16 weeks
Measure: Number; unit: percentage of particpants in arm
Arm/Group | Antidepressant + Desensitization | Antidepressant + Cognitive Behavioral
Number analyzed (Participants) | 75 | 75
percentage of particpants in arm | 29 | 54

ADVERSE EVENTS:
Arm/Group | Antidepressant + Desensitization | Antidepressant + Cognitive Behavioral
Serious Adverse Events (participants affected / at risk) | 3/75 | 2/75
Other Adverse Events (participants affected / at risk) | 0/75 | 1/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antidepressant + Desensitization (N=75) | Antidepressant + Cognitive Behavioral (N=75)
suicidal ideation and worsening depression (Psychiatric disorders) | 0 | 1 — Psychiatric event
Worsening of known cardiac condition (Cardiac disorders) | 0 | 1 — Medical event requiring hospitalization . Event was not expected and was not related to study meds
Severe vaginal bleeding and pain (Reproductive system and breast disorders) | 1 | 0 — Medical event requiring hospitalization.
Chest pain in a patient with CAD (Cardiac disorders) | 1 | 0 — Medical event requiring hospitalization
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Medical event requiring hospitalization The person experiencing this event had another serious adverse event
Hematoma R side abdomen (Blood and lymphatic system disorders) | 1 | 0 — Medical event requiring hospitalization The person experiencing this event had another SAE event
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antidepressant + Desensitization (N=75) | Antidepressant + Cognitive Behavioral (N=75)
Medically significant event not requiring hospitalization (Injury, poisoning and procedural complications) | 0 | 1 — slipped on street curb and broke wrist

LIMITATIONS AND CAVEATS:
Our results do not inform clinical guidelines for any single antidepressant medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No